CLINICAL TRIAL: NCT05974930
Title: Intravascular ULTRAsound-Guided PCI in Patients With ST-Elevation Myocardial Infarction: the ULTRA-STEMI Trial
Brief Title: Intravascular ULTRAsound-Guided PCI in Patients With ST-Elevation Myocardial Infarction
Acronym: ULTRA-STEMI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Karagiannidis Efstratios, Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: 69589
Record Dates: First submitted 2023-07-16; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: STEMI; Intravascular Imaging; IVUS
Keywords: IVUS; Thrombus; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Aspirated thrombotic samples (in cases with large thrombus burden) will be collected to undergo micro-CT scanning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with STEMI undergoing IVUS-guided primary PCI: The ULTRA-STEMI trial will include consecutive patients with STEMI undergoing IVUS-guided primary PCI. All participants will undergo: IVUS intra-coronary imaging at baseline-, post-intervention and post-optimization. If manual thrombus aspiration is needed, the aspirated thrombotic material will be collected to be micro-CT scanned. Post-PCI iFR will be also performed in each participant. Clinical, angiographic and peri-procedural data will be collected. Each participant will be subject to telephone follow-up at 1, 6 and 12 months.
  Interventions: Device: IVUS imaging for primary PCI guidance

INTERVENTIONS:
Device: IVUS imaging for primary PCI guidance — Eagle Eye Platinum Intravascular ultrasound (IVUS) will be used to assess intra-coronary plaque, thrombus or stenosis in patients with STEMI. The device is FDA- and EMA-approved and routinely used in clinical practice. Quantitative and qualitative IVUS parameters will be collected and recorded for all participants to be correlated with clinical, imaging and angiographic outcomes of interest.

SUMMARY:
The main goal of the ULTRA-STEMI trial is to investigate the prognostic impact of IVUS-guided PCI in patients with STEMI and correlate IVUS measurements with clinical, procedural, imaging and follow-up outcomes of interest.

Study participants will undergo primary PCI as per standardized procedures; IVUS will be performed at baseline, post-intervention and post-optimization. Manual thrombus aspiration will be performed according to clinical indications. The aspirated thrombi will be collected and scanned with micro-computed tomography (micro-CT). Also, angiographic and peri-procedural data will be gathered. Post-PCI instantaneous wave-free ratio (IFR) will also be performed to assess the severity of the residual coronary-artery stenosis, if any. All patients will be followed up for at least12 months for the adjudication of major adverse cardiovascular events.

DETAILED DESCRIPTION:
The ULTRA-STEMI trial is a prospective investigator-initiated single-centre single-arm observational cohort study aiming to enroll 80 consecutive patients presenting with ST-segment elevation myocardial infarction (STEMI) and undergoing IVUS-guided primary PCI. IVUS will be performed at baseline, post-intervention and post-optimization. Baseline tissue characterization includes the morphological description of culprit lesion plaque and thrombus characteristics as assessed with IVUS. In patients with large thrombus burden, manual thrombus aspiration will be performed according to clinical indications. The aspirated thrombi will be collected and scanned with micro-computed tomography (micro-CT) to correlate IVUS measurements with micro-CT thrombus quantification. Also, angiographic data will be gathered to correlate IVUS measurements with pre-and post-PCI angiographic information. Post-PCI instantaneous wave-free ratio (IFR) will also be performed to assess the severity of the residual coronary-artery stenosis, if any. All patients will be followed up for at least 12 months for the adjudication of major adverse cardiovascular events.The primary endpoint will be target vessel failure at 12 months (defined as a composite of cardiac death, target vessel myocardial infarction and clinically driven target vessel revascularization). The secondary outcomes of interest will be: radiation exposure, contrast use and kidney function effects. Other endpoints include clinical and angiographic outcomes along with post-PCI IVUS, iFR and micro-CT findings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute STEMI undergoing primary PCI within 12 hours of symptom onset according to the 4th universal definition of myocardial infarction.
2. Age >18 years
3. Individuals willing to voluntarily sign the consent and data protection forms before their inclusion in the clinical study.

Exclusion Criteria:

1. Patients presenting with cardiogenic shock
2. Patients with a known contraindication for primary PCI
3. Pregnancy
4. Presentation ≥12 hours after symptom onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting with STEMI undergoing primary PCI for a native coronary artery culprit lesion will undergo IVUS (at baseline, post-intervention and post-optimization) and post-PCI iFR.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of "Target vessel failure" at 12 months of follow-up in association with IVUS measurements | 2 years
  Follow-up will be obtained using online patient-reported outcome measurements by email or standardized telephone calls at 30 days, 6 months and 12 months after the procedure. Primary follow-up outcome of interest is the composite endpoint of target vessel failure (cardiac death, new-onset heart failure, target vessel myocardial infarction, clinically driven target vessel revascularization or target lesion revascularization).
All-cause mortality at 12 months of follow-up in association with IVUS measurements | 2 years
  Co-primary study outcome will be the investigation of all-cause mortality (i.e., death from any cause) after hospitalization and during follow-up.

SECONDARY OUTCOMES:
In-hospital (post-PCI) adverse events in association with IVUS measurements | 2 years
  The composite endpoint of in-hospital (post-PCI) adverse events includes: cardiac tamponade, need for CABG, shock, in-hospital mortality, acute kidney failure, bleeding, stroke.
Pre-procedural angiographic outcomes in association with IVUS measurements | 2 years
  Pre-procedural Thrombolysis in myocardial infarction (TIMI) flow, thrombus burden classification, culprit vessel, number of diseased vessels, and the SYNergy between percutaneous intervention with TAXus DES and cardiac surgery (SYNTAX) score will be recorded and associated with pre-procedural IVUS measurements. Higher SYNTAX score and lower TIMI flow represent greater obstruction in the diseased vessels.
Post-procedural angiographic outcomes in association with IVUS measurements | 2 years
  Post-procedural TIMI flow, angiographically evident residual thrombus, no-reflow phenomenon, myocardial blush grade, and distal embolization will be recorded and associated with IVUS measurements.
Post-PCI iFR measurement in association with IVUS measurements | 2 years
  iFR=ratio of distal coronary pressure (Pd) to the aortic pressure (Pa) during an isolated period during diastole.
Microtomographic thrombus volume in association with IVUS measurements | 2 years
  Micro-CT derived volume of the extracted thrombotic material will be correlated with IVUS measurements.
Microtomographic thrombus porosity in association with IVUS measurements | 2 years
  Micro-CT derived porosity of the extracted thrombotic material will be correlated with IVUS measurements.
Microtomographic thrombus density in association with IVUS measurements | 2 years
  Micro-CT derived density of the extracted thrombotic material will be correlated with IVUS measurements.
Νumber and type of stents in association with IVUS measurements | 2 years
  Νumber and type of stents used will be recorded and associated with IVUS measurements.
Stent length and diameter in association with IVUS measurements | 2 years
  Stent length and diameter will be recorded and associated with IVUS measurements.
Contrast volume in association with IVUS measurements | 2 years
  Volume of the contrast used will be recorded and associated with IVUS measurements.
Radiation dose in association with IVUS measurements | 2 years
  Peri-procedural radiation dose will be recorded and associated with IVUS measurements.
Procedural duration in association with IVUS measurements | 2 years
  Procedural duration will be recorded and associated with IVUS measurements.
Post-PCI stent underexpansion, deformation or malapposition in association with baseline IVUS measurements | 2 years
  Stent underexpansion, deformation or malapposition (yes/no) will be recorded and associated with baseline IVUS measurements.
Post-PCI edge dissection in association with baseline IVUS measurements | 2 years
  Edge dissection (yes/no) will be recorded and associated with baseline IVUS measurements.
Post-PCI high plaque burden at stent edges, residual focal lesions or tissue protrusion through the stent struts in association with baseline IVUS measurements | 2 years
  High plaque burden at stent edges, residual focal lesions or tissue protrusion through the stent struts (yes/no) will be recorded and associated with baseline IVUS measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Kassimis, MD, PhD, Principal Investigator — 2ND Cardiology Department, Hippokrateion General Hospital of Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Groenland FTW, Mahmoud KD, Neleman T, Ziedses des Plantes AC, Scoccia A, Ligthart J, Witberg KT, Nuis RJ, den Dekker WK, Wilschut JM, Diletti R, Zijlstra F, Kardys I, Cummins P, Van Mieghem NM, Daemen J. Tissue characterisation and primary percutaneous coronary intervention guidance using intravascular ultrasound: rationale and design of the SPECTRUM study. Open Heart. 2022 Apr;9(1):e001955. doi: 10.1136/openhrt-2021-001955. PMID 35437257
- [Background] Karagiannidis E, Papazoglou AS, Sofidis G, Chatzinikolaou E, Keklikoglou K, Panteris E, Kartas A, Stalikas N, Zegkos T, Girtovitis F, Moysidis DV, Stefanopoulos L, Koupidis K, Hadjimiltiades S, Giannakoulas G, Arvanitidis C, Michaelson JS, Karvounis H, Sianos G. Micro-CT-Based Quantification of Extracted Thrombus Burden Characteristics and Association With Angiographic Outcomes in Patients With ST-Elevation Myocardial Infarction: The QUEST-STEMI Study. Front Cardiovasc Med. 2021 Apr 21;8:646064. doi: 10.3389/fcvm.2021.646064. eCollection 2021. PMID 33969012
- [Background] Didagelos M, Pagiantza A, Zegkos T, Zarra K, Angelopoulos V, Kouparanis A, Peteinidou E, Kassimis G, Karvounis H, Ziakas A. Low Molecular Weight Heparin in Improving RAO After Transradial Coronary Catheterization: The LOW-RAO Randomized Study. JACC Cardiovasc Interv. 2022 Aug 22;15(16):1686-1688. doi: 10.1016/j.jcin.2022.05.047. Epub 2022 Jul 27. No abstract available. PMID 35981848